CLINICAL TRIAL: NCT01258634
Title: A Pilot Study of Pre-Operative Treatment of Newly-Diagnosed, Surgically-Resectable Osteosarcoma With Doxorubicin, Ifosfamide, Etoposide, and Cisplatin With Early Metabolic Assessment of Response
Brief Title: A Study of Pre-Operative Treatment of Newly-Diagnosed, Surgically-Resectable Osteosarcoma With Doxorubicin, Ifosfamide, Etoposide, and Cisplatin With Early Metabolic Assessment of Response
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI no longer affiliated with institution; only 2 subjects enrolled
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-186-B
Record Dates: First submitted 2010-09-30; First posted 2010-12-13 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Osteosarcoma; Lung Metastases
Keywords: Osteosarcoma; Surgically Resectable High Grade Osteosarcoma; Lung Metastases Only
MeSH Terms: conditions — Osteosarcoma | interventions — Dexrazoxane; Doxorubicin; Cisplatin; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Etoposide; Ifosfamide; Mesna; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pre-op treatment (Other)
  Interventions: Drug: Dexrazoxane; Drug: Doxorubicin; Drug: Cisplatin; Drug: G-CSF; Drug: PEG-filgrastim; Drug: Etoposide; Drug: Ifosfamide; Drug: Mesna; Drug: Leucovorin

INTERVENTIONS:
Drug: Dexrazoxane — Preoperative Chemotherapy Courses 1, 2, 3, 4: 750mg/m2; IV over 15 minutes on day 1
  Postoperative Chemotherapy for Good Responders Courses 1 and 2: 750mg/m2 IV over 15 minutes on Day 1
  Postoperative Chemotherapy for Poor Responders Courses 2 and 4: 750mg/m2 IV over 15 minutes on Day 1
Drug: Doxorubicin — Preoperative Chemotherapy Courses 1 and 3: 75mg/m2; IV push day 1 Courses 2 and 4: 75mg/m2; IV push day 1, hour 0
  Postoperative Chemotherapy for Good Responders Course 1: 75mg/m2; IV push day 1 Course 2: 75mg/m2; IV push day 1, hour 0
  Postoperative Chemotherapy for Poor Responders Course 2: 75mg/m2; IV push day 1 Course 4: 75mg/m2; IV push day 1, hour 0
Drug: Cisplatin — Preoperative Chemotherapy Courses 1 and 3: 60mg/m2 daily x 2 days, in 1000 ml D5W NS + 10g/m2 mannitol
  Postoperative Chemotherapy for Good Responders Courses 1 and 2: 60mg/m2 daily x 2 days, in 1000 ml D5W NS + 10g/m2 mannitol
  Postoperative Chemotherapy for Poor Responders:
  Course 2: 60mg/m2 daily x 2 days, in 1000 ml D5W NS + 10g/m2 mannitol
Drug: G-CSF — Preoperative Chemotherapy Courses 1, 2, 3, and 4: 5mcg/Kg; IV/SQ starting 24 hours after chemotherapy until WBC >10,000
  Postoperative Chemotherapy for Good Responders Courses 1, 2, and 3: 5mcg/Kg; IV/SQ starting 24 hours after chemotherapy until WBC >10,000
  Postoperative Chemotherapy for Poor Responders Courses 2, 4, and 5: 5mcg/Kg; IV/SQ starting 24 hours after chemotherapy until WBC >10,000
Drug: PEG-filgrastim — Preoperative Chemotherapy Courses 1, 2, 3, and 4: 6mg; SQ starting 24 hours after chemotherapy
  Postoperative Chemotherapy for Good Responders Courses 1, 2, and 3: 6mg; SQ starting 24 hours after chemotherapy
  Postoperative Chemotherapy for Poor Responders Courses 2 and 4: 6mg; SQ starting 24 hours after chemotherapy
Drug: Etoposide — Preoperative Chemotherapy Courses 2 and 4: 50mg/m2 on days 1, 2, 3, 4
  Postoperative Chemotherapy for Good Responders Course 2: 50mg/m2 on days 1, 2, 3, 4 Course 3: 50mg/m2 on days, 1, 2, 3, 4 Hour 0-1
  Postoperative Chemotherapy for Poor Responders Course 4: 50mg/m2 on days 1, 2, 3, 4 Course 5: 50mg/m2 on days 1, 2, 3, 4
Drug: Ifosfamide — Preoperative Chemotherapy Courses 2 and 4: 3g/m2; IV over 1 hour Days 1, 2, 3, 4
  Postoperative Chemotherapy for Good Responders Course 2: 3g/m2; IV over 1 hour Days 1, 2, 3, 4 Course 3: 3g/m2; IV over 1 hour Days 1, 2, 3, 4
  Postoperative Chemotherapy for Poor Responders Course 4: 3g/m2; IV over 1 hour Days 1, 2, 3, 4 Course 5: 3g/m2; IV over 1 hour Days 1, 2, 3, 4
Drug: Mesna — Preoperative Chemotherapy Courses 2 and 4: 600mg/m2, 1st dose in bag with ifosfamide, 2nd dose IV over 3 hours immediately post ifosfamide infusion, Subsequent doses - hour 5, 8, 11, 14 (IV push)
  Postoperative Chemotherapy for Good Responders Courses 2 and 3: 600mg/m2, 1st dose in bag with ifosfamide, 2nd dose IV over 3 hours immediately post ifosfamide infusion, Subsequent doses - hour 5, 8, 11, 14 (IV push)
  Postoperative Chemotherapy for Poor Responders Courses 4 and 5: 600mg/m2, 1st dose in bag with ifosfamide, 2nd dose IV over 3 hours immediately post ifosfamide infusion, Subsequent doses - hour 5, 8, 11, 14 (IV push)
Drug: Leucovorin — Postoperative Chemotherapy for Poor Responders Courses 1 and 3: 15 mg/m2/dose IV or PO every 6 hours, beginning 24 hours after start of methotrexate infusion and continuing until methotrexate level is <0.1 uM

SUMMARY:
This is a pilot study that will allow investigators to collect data related to early and potentially more accurate response assessments using a chemotherapy protocol that eliminates methotrexate to maximize the dose intensity of doxorubicin. The pilot data will be used to seek funding to more fully address the hypotheses in a multi-institutional, Phase II or Phase III trial. The primary and secondary objectives are as follows:

Primary:

1. To evaluate the feasibility and potential usefulness of measuring early changes in tumor metabolic activity, assessed by Fludeoxyglucose-Positron Emission Tomography (FDG-PET) imaging and alkaline phosphatase activity, as early predictors of histological response rate at 12 weeks in osteosarcoma patients.
2. To explore whether histological response can be assessed by a computer algorithm using virtual microscopic images of pathology material, and whether quantifying necrosis in this way correlates with microscope slide-based review.

Secondary:

1. To gather pilot data on the histological response rate, 3-year event-free survival, and toxicity when children and young adults with resectable osteosarcoma are treated using a chemotherapy regimen of alternating courses of doxorubicin/cisplatin (DC) and doxorubicin/ifosfamide/etoposide (IDE).

All patients will receive 4 courses of preoperative chemotherapy courses. With the exception of high-dose methotrexate, which is given weekly, preoperative and postoperative chemotherapy courses are planned to begin every 21 days.

Patients with good histological response (those patients with > 90% tumor necrosis at time of definitive resection) will receive three postoperative chemotherapy courses. The 1st will consist of doxorubicin, dexrazoxane, cisplatin and Granulocyte-Colony Stimulating Factor (G-CSF)(or Polyethylene Glycol filgrastim). The 2nd course will consist of doxorubicin, dexrazoxane, ifosfamide, MESNA, etoposide, G-CSF (or PEG-filgrastim). The 3rd course will consist of ifosfamide, MESNA, etoposide, G-CSF (or PEG-filgrastrim). The total doxorubicin dose will be 450 mg/m2.

Patients with poor response (those patients with < 90% tumor necrosis found on pathology at time of definitive resection) will receive five postoperative chemotherapy courses. High Dose-Methotrexate will be administered during the 1st and 3rd postoperative chemotherapy courses as 4-weekly and 2-weekly doses, respectively. The 2nd course will consist of doxorubicin, dexrazoxane, cisplatin and G-CSF (or PEG-filgrastim). The 4th course will consist of doxorubicin, dexrazoxane, ifosfamide, Mesna, etoposide, G-CSF (or PEG-filgrastim). The 5th cycle will consist of ifosfamide, Mesna, etoposide, G-CSF (or PEG-filgrastrim). The total doxorubicin dose will be 450 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 2 and 35 years of age at time of diagnosis
* Must have biopsy-proven, high-grade osteosarcoma.
* Patients with metastases are eligible as long as the lung is the only site of metastatic disease.
* The primary tumor and all pulmonary metastases must be deemed to be potentially resectable. There must be a commitment by the surgical team to resect the primary tumor at week 12, and pulmonary nodules at any point, unless the clinical situation indicates these interventions are not in the patient's best interest.
* Patients must have normal laboratory values and cardiac function as defined below:
* Creatinine clearance or radioisotope GFR of > or equal to 70ml/min/1.73 m2 OR

A serum creatinine based on age/gender as follows:

Age Maximum Serum Creatinine (mg/dL) Male Female

1 month to < 6 months 0.4 0.4 6 months to < 1 year 0.5 0.5

1. to < 2 years 0.6 0.6
2. to < 6 years 0.8 0.8

6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

* or equal to 16 years 1.7 1.4

  * Cardiac: Adequate cardiac function is defined as:

Shortening fraction of > or equal to 28% by echocardiogram OR Ejection fraction of > or equal to 50% by radionuclide angiogram

* Hepatic: Adequate liver function is described as:

Total bilirubin of < or equal to 1.5 x upper limit of normal (ULN) for age

* Hematologic function: adequate hematologic function is defined as:

ANC > or equal to 1.5 x 10^9/L and platelet count > or equal to 100 x 10^9/L

* Female patients must have a negative pregnancy test
* Female patients who are lactating must agree to stop breast-feeding.
* Patients must not be known to be HIV positive. Testing for HIV is not mandatory.
* Sexually active patients of childbearing potential must agree to use effective contraception.
* Patients must be able to cooperate fully with all planned protocol therapy.
* Signed informed consent MUST be obtained from patient or parent/legal guardian prior to any study procedures and study entry.

Exclusion Criteria:

* Patients with any low-grade osteosarcoma, post-radiation osteosarcoma, and osteosarcoma associated with Paget's disease are not eligible.
* Patients with metastases other than lung metastases are not eligible.
* Patients may not have received prior chemotherapy.

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Feasibility and usefulness of measuring early changes in tumor metabolic activity. | 6 months after last subject has been enrolled
  The feasibility and potential usefulness of measuring early changes in tumor metabolic activity will be assessed by early Fludeoxyglucose-Positron Emission Tomography imaging and alkaline phosphatase activity.

SECONDARY OUTCOMES:
Gather pilot data on the histological response rate | 3 years after last enrolled subject has completed therapy
  To gather pilot data on the histological response rate when children and young adults with resectable osteosarcoma are treated using a chemotherapy regimen of alternating courses of doxorubicin/cisplatin (DC) and doxorubicin/ifosfamide/etoposide (IDE).
Explore whether histological response can be measured by a computer algorithm | 1 year after last enrolled subject has completed therapy
  To explore whether histological response can be measured by a computer algorithm using virtual microscopic images of pathology material, and whether quantifying necrosis in this way correlates with microscope slide-based review.
Gather pilot data on 3-year event-free survival | 3 years after last subject is enrolled
  To gather pilot data on the 3-year event-free survival when children and young adults with resectable osteosarcoma are treated using a chemotherapy regimen of alternating courses of doxorubicin/cisplatin (DC) and doxorubicin/ifosfamide/etoposide (IDE).
Gather pilot data on toxicity | 3 years after last subject is enrolled on the study.
  To gather pilot data on toxicity when children and young adults with resectable osteosarcoma are treated using a chemotherapy regimen of alternating courses of doxorubicin/cisplatin (DC) and doxorubicin/ifosfamide/etoposide (IDE).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen X. Skapek, MD, Principal Investigator — University of Chicago; Andres Morales, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Department of Pediatrics Hematology/Oncology, Chicago, Illinois, United States